CLINICAL TRIAL: NCT03219164
Title: Randomized, Double-Blind, Phase 3B Trial to Evaluate the Safety and Efficacy of 2 Treatment Regimens of Aztreonam 75 mg Powder and Solvent for Nebulizer Solution / Aztreonam for Inhalation Solution (AZLI) in Pediatric Subjects With Cystic Fibrosis (CF) and New Onset Respiratory Tract Pseudomonas Aeruginosa (PA) Infection/Colonization
Brief Title: Study of Aztreonam for Inhalation in Children With Cystic Fibrosis and New Infection of the Airways by Pseudomonas Aeruginosa Bacteria
Acronym: ALPINE 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early by sponsor due to the challenges and risks introduced by Coronavirus disease 2019 (COVID-19) pandemic.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-205-1850; 2016-002749-42 (EudraCT Number)
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Pseudomonas Aeruginosa Respiratory Tract Infection/Colonization; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Aztreonam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZLI + Placebo (Experimental): 75 mg/ml of aztreonam will be administered thrice daily (TID) for 14 days followed by placebo to match (PTM) aztreonam TID for 14 days.
  Interventions: Drug: AZLI; Drug: Placebo
- AZLI (Experimental): 75 mg/ml of aztreonam will be administered TID for 28 days.
  Interventions: Drug: AZLI

INTERVENTIONS:
Drug: AZLI — Administered via the PARI Altera® Nebulizer System. Participants < 2 years will receive via the SmartMask® Baby, 2 to < 6 years via the SmartMask Kids® and > 6 years via the nebulizer mouthpiece.
  Other Names: Cayston®; Aztreonam
Drug: Placebo — Administered via the PARI Altera® Nebulizer System. Participants < 2 years will receive via the SmartMask® Baby, 2 to < 6 years via the SmartMask Kids® and > 6 years via the nebulizer mouthpiece.
  Arms: AZLI + Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of a 14-day course versus a 28-day course of aztreonam for inhalation solution (AZLI) in pediatric participants with new onset Pseudomonas aeruginosa respiratory tract infection or colonization.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of cystic fibrosis (CF) as determined by the 2008 CF Consensus Conference criteria: Sweat chloride level ≥ 60 milliequivalents per liter (mEq/L) by quantitative pilocarpine iontophoresis; or a genotype with 2 identifiable mutations consistent with CF; or an abnormal nasal transepithelial potential difference (NPD), and 1 or more clinical features consistent with CF
* Documented new onset of positive respiratory tract culture for PA within 30 days of screening defined as either first lifetime documented PA-positive culture, or PA recovered after at least a 2-year history of PA-negative respiratory cultures (at least 2 cultures per year)
* Forced expiratory volume in one second (FEV1) ≥ 80% predicted (for subjects ≥ 6 years of age who can reliably perform spirometry assessments)
* Clinically stable with no evidence of acute significant respiratory symptoms that would require administration of intravenous (IV) antipseudomonal antibiotics, oxygen supplementation, or hospitalization

Key Exclusion Criteria:

* Use of IV or inhaled antipseudomonal antibiotics within 2 years of screening
* Use of oral antipseudomonal antibiotics for a respiratory event within 30 days of study entry (screening visit)
* History of intolerance to inhaled short acting β2 agonists
* History of lung transplantation
* Current requirement for daily continuous oxygen supplementation or requirement of more than 2 L/minute at night
* Hospitalization for a respiratory event within 30 days prior to screening
* Changes in bronchodilator, corticosteroid, dornase alfa, or hypertonic saline medications within 7 days prior to screening.
* Significant changes (per investigators discretion) in physiotherapy technique or schedule within 7 days prior to screening
* Abnormal renal or hepatic function results at most recent test within the previous 12 months, defined as Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times upper limit of normal (ULN), or Serum creatinine > 2 times ULN for age
* Presence of a condition or abnormality that would compromise the subject's safety or the quality of the study data, in the opinion of the Investigator
* Known hypersensitivity to aztreonam, its metabolites, or formulation excipients in AZLI
* Respiratory cultures performed within 24 months prior to screening that are positive for ANY Burkholderia spp. or Non-tuberculous mycobacteria (NTM)

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 149 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (53):
- United States (12):
  - University of California San Francisco (UCSF) - Benioff Children's Hospital, San Francisco, California
  - Children's National Health System, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - Ann & Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Corner Children's Hospital, Chicago, Illinois
  - University of Mississippi Medical center, Jackson, Mississippi
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - USC Department of Pediatrics/Division of Pediatric Pulmonology, Columbia, South Carolina
  - Cook Children's Medical Center, Fort Worth, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
- Austria (2):
  - Medizinische Universitat Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
- Belgium (2):
  - Hopital Universitaire des Enfants Reine Fabiola, Brussels
  - UZ Antwerpen, Edegem
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
- France (3):
  - Hopital des enfants - GH Pellegrin, Bordeaux
  - CHU Grenoble Alpes, Grenoble
  - Hopital Robert Debre APHP, Paris
- Germany (2):
  - Universitatsklinikum Essen, Essen
  - Stadtisches Krankenhaus Kiel, Kiel
- General Hospital of Thessaloniki,3rd Dept of Pediatrics, Thessaloniki, Greece
- Israel (4):
  - Rambam Health Corporation, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (6):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Fondazione IRCCS ca Granda, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Policlinico Umberto - Universita La Sapienza di Roma, Roma
  - Ospedale Pediatrico Bambino Gesu, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- VU University Medical Center, Amsterdam, Netherlands
- Spain (7):
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario, Valencia
- United Kingdom (11):
  - NHS Grampian, Aberdeen
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Royal Devon and Exeter Foundation NHS Trust, Exeter
  - University Hospitals of Leicester NHS trust, Leicester
  - Barts and the London Children's Hospital, London
  - Kings College Hospital NHS foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Sheffield Children's Hospital NHS Trust, Sheffield
  - Southampton University Hospitals NHS trust, Southampton General Hospital, Southampton
  - University Hospitals of North Midlands NHS trust Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Derived] Gilchrist FJ, Bui S, Gartner S, McColley SA, Tiddens H, Ruiz G, Stehling F, Alani M, Gurtovaya O, Bresnik M, Watkins TR, Frankovic B, Skov M; ALPINE2 study investigators. ALPINE2: Efficacy and safety of 14-day vs 28-day inhaled aztreonam for Pa eradication in children with cystic fibrosis. J Cyst Fibros. 2024 Jan;23(1):80-86. doi: 10.1016/j.jcf.2023.06.008. Epub 2023 Jul 15. PMID 37455237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe, Israel, and the United States. The first participant was screened on 28 November 2017. The last study visit occurred on 23 September 2021.
Pre-assignment Details: 149 participants were screened.
Groups:
- AZLI 14 Days + Placebo 14 Days: 75 milligrams per milliliter (mg/ml) of aztreonam was administered thrice daily (TID) for 14 days followed by placebo to match (PTM) aztreonam TID for 14 days, both aztreonam and PTM aztreonam were delivered via the PARI Altera® Nebulizer System. Participants below 2 years received aztreonam for inhalation solution (AZLI) and PTM aztreonam via the SmartMask® Baby, 2 to below 6 years via the SmartMask Kids® and above 6 years via the nebulizer mouthpiece.
- AZLI 28 Days: 75 mg/ml of aztreonam was administered TID for 28 days via the PARI Altera® Nebulizer System. Participants below 2 years received AZLI via the SmartMask® Baby, 2 to below 6 years via the SmartMask Kids® and above 6 years via the nebulizer mouthpiece.
Period: Overall Study
Arm/Group | AZLI 14 Days + Placebo 14 Days | AZLI 28 Days
Started | 74 | 75
Completed | 49 | 57
Not Completed | 25 | 18
Not completed — Study Terminated by Sponsor | 16 | 12
Not completed — Withdrew Consent by Parent/Guardian | 5 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrew Assent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were randomized and received at least one dose of study drug.
Groups:
- AZLI 14 Days + Placebo 14 Days: 75 mg/ml of aztreonam was administered TID for 14 days followed by PTM aztreonam TID for 14 days, both aztreonam and PTM aztreonam were delivered via the PARI Altera® Nebulizer System. Participants below 2 years received AZLI and PTM aztreonam via the SmartMask® Baby, 2 to below 6 years via the SmartMask Kids® and above 6 years via the nebulizer mouthpiece.
- Total: Total of all reporting groups
Arm/Group | AZLI 14 Days + Placebo 14 Days | AZLI 28 Days | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.3 (5.34) | 6.5 (4.91) | 6.9 (5.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 39 | 42 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = collection of ethnicity information not allowed by local regulations.
  Participants
    Ethnicity: Not Hispanic or Latino | 66 | 65 | 131
    Ethnicity: Hispanic or Latino | 8 | 9 | 17
    Ethnicity: Not Permitted | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 1 | 1 | 2
  Race: Black or African American | 1 | 0 | 1
  Race: White | 69 | 73 | 142
  Race: Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 17 | 33
  United States | 16 | 16 | 32
  Spain | 6 | 14 | 20
  Italy | 8 | 4 | 12
  France | 6 | 5 | 11
  Denmark | 4 | 5 | 9
  Israel | 4 | 4 | 8
  Austria | 4 | 3 | 7
  Germany | 4 | 3 | 7
  Greece | 3 | 1 | 4
  Belgium | 3 | 0 | 3
  Netherlands | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pseudomonas Aeruginosa (PA)-Negative Cultures Through 28 Days Post-Treatment in the 14-Day Treatment Group vs 28-Day Treatment Group
Time Frame: 28 days post treatment (Weeks 4 to 6 for the 14 Day treatment group and Weeks 4 to 8 for the 28 Day treatment group)
Population: Evaluable Analysis Set included participants who completed study drug with at least 75% compliance, did not use any anti-PA antibiotics while on study treatment with AZLI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZLI 14 Days + Placebo 14 Days | AZLI 28 Days
Number analyzed (Participants) | 68 | 71
percentage of participants | 55.9 [43.3 to 67.9] | 63.4 [51.1 to 74.5]
Statistical Analysis 1: Comparison: AZLI 14 Days + Placebo 14 Days vs AZLI 28 Days; Test type: Non-Inferiority — Non-inferiority of the 14-day treatment regimen was claimed if the lower bound of 1-sided 97.5% confidence limit of the treatment difference (14-day course group vs 28-day course group) was above the noninferiority margin of -20%; Difference in percentage = -8.0, 95% CI 2-sided [-24.6 to 8.6] — The difference in percentage between treatment groups, and the associated 95% CIs were constructed based on stratum-adjusted Mantel-Haenszel method using age as stratification factor

2. Secondary Outcome: Time From Primary Eradication to PA Recurrence Over a 108-Week Post-Treatment Follow-up Period
Description: The primary eradication was achieved when all cultures through 28 days post AZLI treatment were PA negative. Recurrence after PA eradication was defined as first positive PA culture result in participant who successfully met primary endpoint and had no PA-positive culture from local lab at Week 4 through Week 6 for AZLI 14 Days group or through Week 8 for AZLI 28 Days group.
Time Frame: Last dose date of AZLI up to Week 112
Population: Participants in the Evaluable Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | AZLI 14 Days + Placebo 14 Days | AZLI 28 Days
Number analyzed (Participants) | 68 | 71
months | 19.3 [10.5 to NA] — Not Available as the calculated percentiles of event rate were not reached. | NA [4.9 to NA] — Not Available as the calculated percentiles of event rate were not reached.

3. Secondary Outcome: Percentage of Participants With PA-negative Cultures Through 28 Days Post-Treatment in the 14-Day Treatment Group vs Historical Pooled Data for PA Eradication at 28 Days Post-Treatment in Participants Treated With Tobramycin Nebulizer Solution (TNS)
Time Frame: 28 days post treatment (Weeks 4 to 6 for the 14 Day treatment group)
Population: AZLI 14 Day treatment group: Evaluable Analysis Set. No data was collected for the AZLI 28 Day treatment group for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | AZLI 14 Days + Placebo 14 Days
Number analyzed (Participants) | 68
percentage of participants | 55.9
Statistical Analysis 1: Comparison: AZLI 14 Days + Placebo 14 Days; Test type: Other; The historical pooled data from published results for the percentage of participants with successful PA eradication at 28 days post-treatment with TNS was estimated to be 77%

4. Secondary Outcome: Time to PA Recurrence for a Sub-Group of Participants Matching the Population in the TNS ELITE Study Over a 108-Week Post-Treatment Follow-up Period
Description: In ELITE study (NCT00391976), participants with cystic fibrosis who had early PA infection received TNS. Published criteria for efficacy analysis population in ELITE study included:
  * Participants must be ≥ 6 months at randomization
  * No history of positive anti-PA antibody (no anti-PA immunoglobulin G [IgG] antibody interpretation at Screening/Baseline) on record
  * Did not use anti-pseudomonal antibiotics through 28 days after completion of active treatment and within 2 years of Screening
  * Non-missing PA culture result at 28 days after last dose of AZLI
  * PA negative through 28 days after completion of active treatment
  * No important protocol deviation related to compliance with study drug administration
  * Documented new onset of positive respiratory tract culture for PA within 30 days of Screening defined as either first lifetime documented PA-positive culture, or PA recovered after at least a 2-year history of PA-negative respiratory cultures (at least 2 cultures per year).
Time Frame: Last dose date of AZLI up to Week 112
Population: ELITE Study Matching Analysis Set included participants from Evaluable Analysis Set (who did not meet evaluability criteria due to < 75% compliance, use of anti-PA antibiotics while on AZLI treatment, missing PA culture result during initial eradication phase) who also satisfied the published criteria for efficacy analysis population in ELITE study.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | AZLI 14 Days + Placebo 14 Days | AZLI 28 Days
Number analyzed (Participants) | 23 | 25
months | 19.3 [10.5 to NA] — Not Available as the calculated percentiles of event rate were not reached. | 15.2 [4.7 to NA] — Not Available as the calculated percentiles of event rate were not reached.

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 28 days plus 30 days; All-Cause Mortality: Randomization up to 112 weeks
Description: Adverse Events: Safety Analysis Set included participants who were randomized and received at least one dose of study drug.
  All-Cause Mortality: Intent-To-Treat Analysis Set included all participants who were randomized in the study.
Arm/Group | AZLI 14 Days + Placebo 14 Days | AZLI 28 Days
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 5/74 | 4/75
Other Adverse Events (participants affected / at risk) | 28/74 | 22/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI 14 Days + Placebo 14 Days (N=74) | AZLI 28 Days (N=75)
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Pseudomonas test positive (Investigations) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI 14 Days + Placebo 14 Days (N=74) | AZLI 28 Days (N=75)
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Pyrexia (General disorders) | 4 | 6
Influenza (Infections and infestations) | 1 | 5
Rhinitis (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 11

LIMITATIONS AND CAVEATS:
The study was terminated early due to Coronavirus disease 2019 (COVID-19) pandemic. At the time of study termination, all evaluable participants completed the initial eradication period and provided data for the primary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03219164/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT03219164/SAP_001.pdf